CLINICAL TRIAL: NCT04272658
Title: Interest in PET/CT Whole-body Dynamic Acquisition at FDG to Differentiate Progression/Pseudo Progression of Metastatic Melanoma Under Immunotherapy
Brief Title: PET/CT Whole-body Dynamic Acquisition at FDG to Metastatic Melanoma Under Immunotherapy
Acronym: IMMUNOPET2
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC19.0194 (IMMUNO-PET2)
Record Dates: First submitted 2020-01-20; First posted 2020-02-17 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2023-12

CONDITIONS: Metastatic Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- value of 4D body-to-whole dynamic acquisition in FDG: differentiate pseudo-progression / progression during the first therapeutic assessment by FDG PET / CT (PET1) using data from the 4D whole-body dynamic acquisition, without having to re-evaluate closely. during a PET1 'this "unconfirmed progression" after 2 new treatment cures of immune checkpoint inhibitors in metastatic melanoma
  Interventions: Diagnostic Test: value of 4D body-to-whole dynamic acquisition in FDG

INTERVENTIONS:
Diagnostic Test: value of 4D body-to-whole dynamic acquisition in FDG — differentiate pseudo-progression / progression during the first therapeutic assessment by FDG PET / CT (PET1) using data from the 4D whole-body dynamic acquisition, without having to re-evaluate closely. during a PET1 'this "unconfirmed progression" after 2 new treatment cures of ICI

SUMMARY:
The value of 4D body-to-whole dynamic acquisition in FDG PET / CT to differentiate progression / pseudo-progression during the first therapeutic assessment (PET1) of metastatic melanoma treated with immune checkpoint inhibitors (ICI)to predict the progression of the disease..

ELIGIBILITY:
Inclusion Criteria:

* Patient old ≥ 18 years
* With metastatic melanoma
* Treated with anti-PD1 : Nivolumab or Pembrolizumab or Combo IPI-Nivo
* Having formulated a non-opposition

Exclusion Criteria:

* - Minor patient < 18 years
* Pregnancy or breastfeeding
* Other type of tumor than metastatic melanoma
* Non-eligibility for the examination
* Refusal of participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic melanoma treated with immune checkpoint inhibitors (ICI) and do 4D body-to-whole dynamic acquisition in FDG PET / CT to differentiate progression / pseudo-progression
Sampling Method: Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2020-06-26 (Actual); Primary Completion 2026-06-26 (Estimated); Study Completion 2026-06-26 (Estimated)

PRIMARY OUTCOMES:
Values of the Ki absorption coefficient resulting from a FDG PET / CT full-body 4D dynamic acquisition to differentiate the pseudo-progression / progression of metastatic melanoma treated with ICI | 5 years

SECONDARY OUTCOMES:
Correlation between the Ki lesion values derived from PET1 and the quantitative parameters resulting from PET0 histological specifications of the tumors (% PD-L1, T-CD8 infiltration, PTEN status) to differentiate pseudo-progression / progression. | 5 years
Correlation between the Ki lesional values resulting from the 4D acquisition of the PET / CT from PET1 and PET0 the biological parameters (LDH, leucocytes, neutrophils) to differentiate pseudo-progression / progression | 5 years
Correlation between the Ki lesion values resulting from the 4D acquisition of FDG PET / CT for PET1 and the quantitative parameters resulting from PET0 to differentiate pseudo-progression / progression | 5 years
Correlation between lesional Ki values resulting from the 4D acquisition of FDG PET / CT for from PET1 and the quantitative parameters resulting from PET0 ICI- related adverse effect to differentiate pseudo-progression / progression | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ronan ABGRAL, MD-PhD, Principal Investigator — Nuclear Medecine
Locations (1):
- Hospital University ff Brest, Brest, Finistere, France

IPD SHARING:
Plan to Share IPD: No